CLINICAL TRIAL: NCT03816124
Title: The Effect of Radiofrequency Ablation of Genicular Nerves on Postural Stability in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2018.663
Record Dates: First submitted 2018-12-03; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Patients with knee osteoarthritis with Kellgren-Lawrance scale stage 3-4 will receive radiofrequency ablation to their genicular nerves and will be evaluated before treatment, 3 weeks and 3 months after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genicular RF (Experimental): Patients who will receive genicular radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — radiofrequency ablation of the genicular nerves

SUMMARY:
In advanced knee osteoarthritis, postural stability is also disturbed. There are some concerns about performing radiofrequency ablation to genicular nerves since this may further decrease the postural stability of the patient. The aim of this study is to see if application of genicular radiofrequency causes a significant change in postural stability.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 and 4 knee osteoarthritis according to Kellgren-Lawrance scale
* Knee pain more than 3 months

Exclusion Criteria:

* Neurological diseases such as polyneuropathies
* Presence of severe psychiatric disorders
* Hemodynamic instability
* History of any surgery from the knee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 3 weeks and 3 months after the intervention
  The change of pain will be evaluated with 10 cm visual analogue scale will be applied to the patients, 0 being no pain while 10 being intolerable pain

SECONDARY OUTCOMES:
Postural stability | 3 weeks and 3 months after the treatment
  The change of weight bearing indexes of both feet will be measured
WOMAC | 3 weeks and 3 months after the treatment
  Western Ontario & McMaster Universities Osteoarthritis Index

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No